CLINICAL TRIAL: NCT01051518
Title: Clinical Evaluation of Percutaneous Implantation of the CoreValve Aortic Valve Prosthesis. Safety and Performance Study on Patients at High Risk for Surgical Valve Replacement (18Fr Safety and Efficacy Study)
Brief Title: Clinical Evaluation of Percutaneous Implantation of the Medtronic CoreValve Aortic Valve Prosthesis (18Fr-Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COR-2006-02
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CoreValve (Experimental)
  Interventions: Device: Medtronic CoreValve System

INTERVENTIONS:
Device: Medtronic CoreValve System — Transcatheter Aortic Valve
  Other Names: Medtronic CoreValve Trancatheter Aortic Valve; Medtronic CoreValve Percutaneous Aortic Valve

SUMMARY:
The investigation concerns a prospective, multicenter, single arm safety and performance study evaluating the Medtronic CoreValve system. Approximately 120 patients presenting with symptomatic aortic native valve stenosis necessitating valve replacement which are considered poor surgical candidates, with a high surgical risk, as attested to by both the surgeon and the cardiologist are recruited in the study.

Safety and performance will be evaluated at discharge and at 30 days post-procedure. Valve performance and placement will be followed up at 3 and 6 months post-procedure. Further long-term patient follow-up visits will be performed at 12, 24, 36 and 48 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Native aortic valve disease, defined as valve stenosis with an aortic valve area <1cm² (<0.6cm2/m2) as determined by echocardiographic measure,
* ≥ 75 years, or
* Surgical risk calculated with logistic EuroSCORE ≥ 15 %, or
* One or two (but not more than 2) of the following complicating factors:

  1. Cirrhosis of the liver (Child class A or B),
  2. Pulmonary insufficiency : Forced expiratory volume in one second (FEV1) < 1 liter,
  3. Previous cardiac surgery (Coronary artery bypass grafting (CABG), valvular surgery),
  4. Pulmonary hypertension > 60 mmHg and high risk of cardiac surgery other than valve replacement,
  5. Porcelain aorta
  6. Recurrent pulmonary embolus,
  7. Right ventricular insufficiency,
  8. Thoracic burning sequelae contraindicating open chest surgery,
  9. History of mediastinum radiotherapy,
  10. Severe connective tissue disease resulting in a contraindication to surgery,
  11. Cachexia (BMI ≤ 18 kg/m²),
* Aortic valve annulus diameter is ≥ 20 mm and ≤ 27 mm as determined by echocardiographic measure,
* Ascending aorta diameter £ 45 mm at the sino-tubular junction, and
* Signed Informed Consent.

Exclusion Criteria:

* Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, Nitinol, or sensitivity to contrast media which cannot be adequately pre-medicated,
* Any sepsis, including active endocarditis,
* Recent myocardial infarction (< 30 days),
* Percutaneous coronary or vascular intervention within 15 days prior to the study procedure, or scheduled during or within 30 days after the study procedure,
* Any left ventricular or atrial thrombus diagnosed by echocardiography,
* Uncontrolled atrial fibrillation (heart rate greater than 100 bpm),
* Mitral or tricuspid valvular insufficiency ( > grade II),
* Previous aortic valve replacement (mechanical valve OR stented bioprosthetic valve),
* Any condition considered as contraindication for extracorporeal assistance,
* Evolutive or recent CVA (cerebro vascular accident),
* Poly arterial patients with either:

  1. Femoral, iliac or aortic vascular condition (e.g. stenosis, tortuosity), that make insertion and endovascular access to the aortic valve impossible, or
  2. Symptomatic carotid or vertebral arteries narrowing (> 70%) disease, or
  3. Abdominal or thoracic aortic aneurysm,
* Bleeding diathesis or coagulopathy, or patient who will refuse blood transfusion,
* Evolutive disease with life expectancy less than one year,
* Creatinine clearance < 20 ml/min,
* Pregnancy, and
* Enrolled in another investigational study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 126 (Actual)
Dates: Start 2006-05; Primary Completion 2009-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Grube, Prof. Dr., Principal Investigator — Helios Heart Center Siegburg, Germany; G. Schuler, Prof. Dr., Principal Investigator — Herzzentrum Universitat Leipzig, Germany; R. Bonan, Dr., Principal Investigator — Institut de Cardiologie de Montreal, Canada; J. Kovac, Dr., Principal Investigator — Glenfield Hospital Leicester, UK; P. Serruys, Prof. Dr., Principal Investigator — Erasmus MC Rotterdam, Netherlands; M. Labinaz, Dr., Principal Investigator — University of Ottawa Heart Institute, Canada; P den Heijer, Dr., Principal Investigator — Amphia Hospital Breda, Netherlands; M Mullen, Dr., Principal Investigator — Royal Brompton & Harefield NHS Trust London, UK; W. Tymchak, Dr., Principal Investigator — University of Alberta Hospital, Canada
Locations (9):
- Canada (3):
  - University of Alberta Hospital, Edmonton
  - Institut de Cardiologie de Montreal, Montreal
  - University of Ottawa Heart Institute, Ottawa
- Germany (2):
  - Herzzentrum Leipzig GmbH, Leipzig
  - HELIOS Heart Center Siegburg, Siegburg
- Netherlands (2):
  - Amphia Hospital, Breda
  - Erasmus MC, Rotterdam
- United Kingdom (2):
  - Glenfield Hospital, Leicester
  - Royal Brompton & Harefield NHS Trust, London

REFERENCES:
- See also: Related Info — http://www.medtronic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nine sites from Western Europe and Canada enrolled 126 subjects between May 2006 and November 2008.
Pre-assignment Details: Of 126 subjects enrolled, 124 were implanted with the CoreValve aortic valve.
Groups:
- Overall Study: All enrolled subjects for whom the procedure of percutaneous implantation of the Medtronic CoreValve aortic valve prosthesis was started.
Period: Overall Study
Arm/Group | Overall Study
Started | 126
Completed | 53
Not Completed | 73

BASELINE CHARACTERISTICS:
Population: Overall study population was divided in high and moderate risk groups based on the risk of operative mortality. The risk classification was performed by 2 independent cardiovascular surgeons who were blinded to procedural details and outcomes but were provided with the baseline logistic EuroSCORE, baseline data and available source documentation.
Groups:
- High Risk: Subjects with a high risk of operative mortality.
- Moderate Risk: Subjects with a moderate risk of operative mortality.
- Total: Total of all reporting groups
Arm/Group | High Risk | Moderate Risk | Total
Number analyzed (Participants) | 72 | 54 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 81.3 (7.2) | 83.8 (4.9) | 82.4 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 72
  Male | 34 | 20 | 54
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 17 | 14 | 31
  Netherlands | 7 | 9 | 16
  United Kingdom | 9 | 9 | 18
  Germany | 39 | 22 | 61
EuroSCORE [Mean (Standard Deviation); unit: Percent of predicted operative mortality] — Measure Description: EuroSCORE: European System for Cardiac Operative Risk Evaluation. Is a measure for predicted operative mortality for patients undergoing cardiac surgery. If a risk factor is present, a weight/number is assigned. The weights are added to give an approximate percent of predicted mortality. The resulting scores are provided on a scale ranging from 0% (no risk at all) to 100% (inoperable) .
  Percent of predicted operative mortality | 28.9 (14.5) | 16.1 (8.5) | 23.4 (13.8)
NYHA [Count of Participants; unit: Participants] — New York Heart Association (NYHA): I) No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea. II) Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea. III) Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea. IV) Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants
    NYHA class I | 2 | 5 | 7
    NYHA class II | 12 | 13 | 25
    NYHA class III | 37 | 31 | 68
    NYHA class IV | 21 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Composite Major Adverse Event (MAE) Free Rate
Description: Percentage of subjects without a composite major adverse event (MAE) at 30 (+ 7) days post-procedure. MAE included all-cause death, non-fatal myocardial infarction, stroke, emergent cardiac re-intervention, cardiac tamponade, non-structural or structural valve dysfunction, cardiogenic shock, endocarditis, TIA, embolism, aortic dissection, access site vessel dissection, vessel perforation, acute vessel occlusion, major bleeding and major vascular injury.
Time Frame: 30 (+7) days post procedure
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Overall Study: All enrolled subjects for whom the procedure for percutaneous implantation of the Medtronic CoreValve aortic valve prosthesis was started.
Arm/Group | High Risk | Moderate Risk | Overall Study
Number analyzed (Participants) | 72 | 54 | 126
Percentage of subjects | 54.2 [42.0 to 66.0] | 48.1 [34.3 to 62.2] | 51.6 [42.5 to 60.6]

2. Secondary Outcome: Composite Technical Device Success
Description: Composite technical success was defined as the percentage of subjects in whom success on all four technical measures of the "Device Functionality Assessment" was achieved and who were adjudicated as having no device failure or malfunction.
  The four measures of the ''Device Functionality Assessment'' were:
  * Load the valve delivery system using the loading system
  * Access the aortic valve with the delivery catheter
  * Deploy the valve accurately across the native aortic valve
  * Remove the intact delivery system
Time Frame: Was assessed during the procedure and completed once the procedure was conlcluded
Population: For two patients in the moderate risk group the composite technical device success could not be calculated because not all measurements required were available.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- High Risk With Complete Device Success Data: Subjects with a high risk of operative mortality with all data available to calculate the composite technical device success
- Moderate Risk With Complete Device Success Data: Subjects with a moderate risk of operative mortality with all data available to calculate the composite technical device success
Arm/Group | High Risk With Complete Device Success Data | Moderate Risk With Complete Device Success Data | Overall Study
Number analyzed (Participants) | 72 | 52 | 124
Percentage of subjects | 84.7 [74.3 to 92.1] | 80.8 [67.5 to 90.4] | 83.1 [75.3 to 89.2]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from date of implantation till 4 years follow up
Groups:
- High Risk; Moderate Risk: Overall study population was divided in high and moderate risk groups based on the risk of operative mortality. The risk classification was performed by 2 independent cardiovascular surgeons who were blinded to procedural details and outcomes but were provided with the baseline logistic EuroSCORE, baseline data and available source documentation.
Arm/Group | High Risk | Moderate Risk
All-Cause Mortality (participants affected / at risk) | 47/72 | 20/54
Serious Adverse Events (participants affected / at risk) | 68/72 | 46/54
Other Adverse Events (participants affected / at risk) | 64/72 | 47/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk (N=72) | Moderate Risk (N=54)
(Blood and lymphatic system disorders) | 9 (11) | 2 (2)
(Cardiac disorders) | 47 (81) | 34 (49)
(Endocrine disorders) | 2 (2) | 0 (0)
(Gastrointestinal disorders) | 14 (14) | 6 (8)
(General disorders) | 18 (21) | 9 (10) — Any other reported adverse events not assosiated with the use of the study device were collected without specyfying a specific adverse event term
(Infections and infestations) | 23 (36) | 9 (11)
(Injury, poisoning and procedural complications) | 11 (12) | 6 (7)
(Investigations) | 1 (1) | 0 (0)
(Metabolism and nutrition disorders) | 4 (4) | 0 (0)
(Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (3)
(Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 0 (0)
(Nervous system disorders) | 17 (20) | 10 (10)
(Product Issues) | 3 (3) | 2 (2)
(Psychiatric disorders) | 2 (2) | 2 (2)
(Renal and urinary disorders) | 12 (13) | 4 (5)
(Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
(Surgical and medical procedures) | 8 (9) | 5 (5)
(Vascular disorders) | 13 (14) | 6 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Risk (N=72) | Moderate Risk (N=54)
(Blood and lymphatic system disorders) | 17 (19) | 16 (18)
(Cardiac disorders) | 32 (40) | 19 (29)
(Congenital, familial and genetic disorders) | 2 (2) | 1 (1)
(Gastrointestinal disorders) | 10 (12) | 7 (8)
(General disorders) | 16 (21) | 11 (15)
(Infections and infestations) | 24 (32) | 21 (26)
(Injury, poisoning and procedural complications) | 7 (8) | 5 (5)
(Investigations) | 6 (6) | 7 (7)
(Metabolism and nutrition disorders) | 3 (3) | 3 (5)
(Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4)
(Nervous system disorders) | 10 (13) | 9 (14)
(Psychiatric disorders) | 2 (2) | 6 (6)
(Renal and urinary disorders) | 17 (20) | 7 (7)
(Reproductive system and breast disorders) | 2 (2) | 0 (0)
(Respiratory, thoracic and mediastinal disorders) | 20 (23) | 12 (18)
(Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
(Surgical and medical procedures) | 3 (6) | 1 (1)
(Vascular disorders) | 23 (32) | 12 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less